CLINICAL TRIAL: NCT06257927
Title: Evaluating the Implementation of a Family Therapy Intervention ("Tuko Pamoja") Delivered Through Sexual and Reproductive Healthcare Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Center for Global Reproductive Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0183
Record Dates: First submitted 2024-01-29; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Family Conflict; Family Dysfunctional; Adolescent Behavior; Child Behavior; Marital Conflict; Domestic Violence; Parent-Child Relations
Keywords: Kenya; Family Therapy
MeSH Terms: conditions — Adolescent Behavior; Child Behavior

STUDY DESIGN:
Intervention Model Description: The study will follow a single case (N of 1) series design. Pre-post changes will be measured, and repeated measures will be administered before, during, and following the intervention to track change over time. The timing of entry into the study and the numbers of repeated measures data points are randomized across families. Data analysis will aim to (a) identify patterns of change over the course of the intervention and (b) relate change trajectories to theorized mechanisms of action.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Tuko Pamoja

INTERVENTIONS:
Behavioral: Tuko Pamoja — Tuko Pamoja, "We are Together" in Kiswahili; This intervention, delivered by lay counselors and through existing community social structures, focuses on improving family relationships and mental health with content derived from evidence-based practices; these include solution-focused family therapy and cognitive behavioral strategies. It is components based, with modules delivered based on need. Tuko Pamoja includes a smart phone component to support psychoeducation components and data collection. The content and structure has been adapted in both content and implementation model based on formative research in this context.

SUMMARY:
This study aims to contribute to the evidence base related to effective interventions for families in low-resource settings who are experiencing conflict and difficulties in relationships that affect child and caregiver well being alike. Results of this study will (a) inform whether a family therapy approach is feasible and promising in communities in and surrounding Kisumu, Kenya and (b) inform how family wellbeing and mental health can be integrated within the sexual reproductive health service points through culturally-valid ways in this context.

Main Objective: To pilot test the implementation of a family therapy intervention (Tuko Pamoja) in collaboration with two sexual and reproductive healthcare settings in Kisumu, Kenya. Specific Objective: To pilot test the Tuko Pamoja family therapy intervention to assess feasibility, acceptability, and preliminary effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Family with self-reported elevated distress (e.g., high levels of conflict) that also has a child/adolescent (ages 8-17) with caregiver-reported emotional or behavioral concerns

Exclusion Criteria:

* Families without reported distress and/or without reported adolescent distress.
* Families with children older than 17 or younger than 8 years of age.
* Families in which primary caregivers or children are living too far outside of the community to participate in treatment.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Family Functioning: Survey Measure | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  30 self-report items developed for the local context based on formative research. Responses are endorsed on a 10-point scale and refer to the past month. One composite score is calculated; higher scores reflect better family functioning. A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Family Functioning: Direct Observation | Baseline and 1 month post-intervention
  A direct observational measure in which families complete standardized video-recorded activities. Behaviors are then coded on multiple domains, including ones related to positive/negative interactions, quality of communication, and problem-solving ability. Primary analyses will be conducted with higher scores indicating better functioning.
Parent-Child Relationship | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Parent-Child Relationship: from standardized scales and locally developed items. Items selected and adapted from: (1) Parental Acceptance and Rejection Questionnaire, (2) Multiple Indicators Cluster Survey: Discipline Module, (3) Discipline Interview, (4) Parent-Adolescent Communication Scale. Each include caregiver and child/adolescent report versions. Caregiver report includes 66 items; Child report includes 60 items. Participants are asked to respond based on the past month. Children report on each caregiver separately.
  For primary analyses, one composite score will be calculated. For follow-up analyses, subsets of items may be analyzed, including those related specifically to harsh treatment/abuse.
  A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Couples Relationship | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Locally-derived items and selected items adapted from standardized scales: Conflict Tactics Scale; Dyadic Adjustment Scale; additional locally-derived items. A total of 52 items are included, referring to both self and spouse behaviors. The majority of items are based on a frequency scale, referring to the past month; some items related to spousal maltreatment assess whether behaviors have ever occurred.
  As a primary outcome, responses across these items will be combined into one score. Follow-up analyses may be conducted using subsets of items to assess relationship quality and harsh treatment separately.
  A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Child / Adolescent Mental Health | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Items locally developed and adapted from standardized measures, including the Youth Self Report (YSR) and the Child Behavior Checklist (CBCL; for caregivers); locally-developed items assessed local terms reflecting symptoms, hope, prosocial behavior, risk behavior, and sense of belongingness. The majority of items reported on a 3-point scale (Not/Never True, Somewhat/Sometimes True, Very/Often True). Caregiver-report on child included 47 items; Child self-report included 56 items. A single composite score will be calculated, with potential follow-up analyses on subsets of items.
  A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.
Caregiver Mental Health | Baseline and 1 month post-intervention; repeated measures pre, during, and post intervention up to 4 weeks
  Locally-developed items and items adapted from subscales of standardized measures, including: Patient Health Questionnaire, General Health Questionnaire. Caregivers self-report on 29 total items. One composite score will be calculated, and potential follow-up analyses may examine subsets of items.
  A subset of these are administered repeatedly pre- and post-intervention as part of the single case series design multiple assessments.

SECONDARY OUTCOMES:
Counselor Implementation Outcomes | Through study completion, approximately 6 months
  This measure will assess feasibility, acceptability, and quality of delivery model.
  Fidelity (Checklists, session transcript analysis) Lay counselor competency (session transcript ratings; Adapted ENACT), including counselor use of community practices (session transcript analysis)
  A composite score will be calculated, and follow-up analyses may examine subsets of items dividing fidelity and competency scores.

CONTACTS AND LOCATIONS:
Overall Officials: Eve S Puffer, PhD, Principal Investigator — Duke University; Megan Huchko, MD, MPH, Principal Investigator — Duke University
Locations (2):
- Kenya (2):
  - Kisumu County Referral Hospital, Kisumu
  - Lumumba Sub-County Hospital, Kisumu

IPD SHARING:
Plan to Share IPD: No